CLINICAL TRIAL: NCT03046433
Title: Children-Adult Asthma Cohort Study in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Children's Hospital (Other)
Collaborators: Shengjing Hospital (Other); Capital Institute of Pediatrics, China (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); China-Japan Friendship Hospital (Other); Ruijin Hospital (Other); Xiangya Hospital of Central South University (Other); Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Kunling Shen, Chief of China National Clinical Research Center for Respiratory Diseases, Beijing Children's Hospital
Other Study IDs: BCHlung008
Record Dates: First submitted 2017-01-25; First posted 2017-02-08 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Asthma in Children
Keywords: children; asthma; China
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a multicenter and prospective cohort study of children diagnosed with asthma. Clinical symptoms and signs, quality of life, blood test, and lung function were detected every three months. FeNO detection, chest imaging, and induced sputum smear were detected when necessary. Biological samples will be collected when recruiting and finishing follow-up.

DETAILED DESCRIPTION:
Asthma is one of the most common chronic diseases all over the world. GINA (Global Initiative for Asthma) reported that nearly 300 million were diagnosed with asthma, while in China even reach to 30 million. In recent years, the prevalence of pediatric asthma and severe cases in China has increased considerably. In 2013, the third national survey carried out in 43 cities in 27 provinces and found that asthma prevalence among children aged 0-14 years old reached to 3.02%, with the highest prevalence in Shanghai (7.57%), while in year of 2000, the rat was 1.09%. However, the research about mechanism, risk factors, individualized prevention and treatment strategy of asthma in China is still not perfect and there is no basic data and multicenter cohort study. Therefore, this multicenter cohort study is conducted, in order to set up a complete database, biobank and long term follow up of Chinese children, and establish foundations for basic research and precise medicine.

Pediatric patients more than or equal to 6 years old diagnosed with asthma will be recruited in this study. After evaluating the baseline, the patients were followed up. Visiting doctors and filling in a questionnaire for every three months, the clinical symptoms, physical examination, will be detected. Chest X ray, blood tests, lung function test and FeNO test would be done when necessary. And, biological samples of blood, urine and throat swab will be collected when recruiting and finishing follow-up. The trial will be completed in 60 months, with 4000 subjects recruited from 8 hospitals.

ELIGIBILITY:
Inclusion Criteria:

1. Age: More than or equal to 6 years old
2. Fulfilling the diagnosis criteria of asthma or cough variant asthma (CVA) based on the guideline of China.
3. The patients cooperated very well with the doctors to perform lung function test.

Asthma is defined as fulfilling followings 1-4 or 4 and 5:

1. History of variable respiratory symptoms: wheezing, shortness of breath, chest tightness, and coughing. Symptoms are often worse at night or upon awakening, and often triggered by exercise, laughter, allergens, or cold air, viral infections.
2. At onset, scattered wheeze in the lungs is heard with prolonged expiratory time.
3. The above symptoms and signs were efficient for anti-asthma, or alleviates voluntarily.
4. Exclusive of other diseases with wheezing, shortness of breath, chest tightness, and coughing.
5. If the manifestation is non-typical, fulfilling one of the followings:

   * Documented airflow limitation：

     1. Positive BD reversibility test: Increase in FEV1 of >12% from baseline, 15 minutes after inhalation of 200-400 μg albuterol;
     2. Significantly increased in lung function after anti-inflammatory treatment;
     3. Increase in FEV1 of >12%, after 4 to 8 weeks of treatment with inhaled corticosteroids and (or) anti-leukotrienes.
   * Positive bronchial challenge test;
   * Excessive variability in twice-daily PEF over 2 weeks: Average daily diurnal PEF variability >13%.

Cough variant asthma (CVA) is defined as fulfilling following:

1. Cough at least 4 weeks without sputum and wheeze, worsening at night or upon awakening;
2. No symptoms of infection, or no effect on long term antibiotic treatment;
3. The symptoms and signs were efficient for anti-asthma treatment;
4. Exclusive of other diseases causing wheeze;
5. Positive exercise challenge test and (or) average daily diurnal PEF variability >13%;
6. Individual or primary, secondary relatives with allergic history, or positive allergen detection.

Exclusion Criteria:

Subject will be excluded if she or he has one of the following:

1. congenital heart disease;
2. heart failure;
3. liver failure or renal insufficiency;
4. kidney disease;
5. connective tissue disease;
6. immunodeficiency;
7. tumor;
8. a history of hypertension or diabetes mellitus.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who was confirmed diagnosis as asthma or cough variant asthma (CVA) at the certain hospitals (sponsor and collaborators)
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Long-term changes on lung function of Chinese children with asthma when treated according to GINA guideline | 60 months

SECONDARY OUTCOMES:
Asthma Quality of Life Questionnaire with Standardized Activities | 3 months
Asthma Control Questionnaire | 3 months
Frequencies of acute attack of asthma in children | 60 months
  Times of acute asthmatic attack will be recorded every year from baseline to 60 months, assessed by questionnaire.
Complications of children with pediatric asthma | 60 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pedersen SE, Hurd SS, Lemanske RF Jr, Becker A, Zar HJ, Sly PD, Soto-Quiroz M, Wong G, Bateman ED; Global Initiative for Asthma. Global strategy for the diagnosis and management of asthma in children 5 years and younger. Pediatr Pulmonol. 2011 Jan;46(1):1-17. doi: 10.1002/ppul.21321. Epub 2010 Oct 20. PMID 20963782
- [Background] Boulet LP, FitzGerald JM, Reddel HK. The revised 2014 GINA strategy report: opportunities for change. Curr Opin Pulm Med. 2015 Jan;21(1):1-7. doi: 10.1097/MCP.0000000000000125. PMID 25405667
- [Background] National Cooperative Group on Childhood Asthma; Institute of Environmental Health and Related Product Safety, Chinese Center for Disease Control and Prevention; Chinese Center for Disease Control and Prevention. [Third nationwide survey of childhood asthma in urban areas of China]. Zhonghua Er Ke Za Zhi. 2013 Oct;51(10):729-35. Chinese. PMID 24406223
- [Background] Subspecialty Group of Respiratory Diseases, Society of Pediatrics, Chinese Medical Association; Editorial Board, Chinese Journal of Pediatrics. [Guideline for the diagnosis and optimal management of asthma in children(2016)]. Zhonghua Er Ke Za Zhi. 2016 Mar;54(3):167-81. doi: 10.3760/cma.j.issn.0578-1310.2016.03.003. No abstract available. Chinese. PMID 26957061